CLINICAL TRIAL: NCT03594656
Title: Effects of Lingzhi on Disease Progression in Patients With Untreated Early Parkinson's Disease: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effects of Lingzhi on Disease Progression in Patients With Untreated Early Parkinson's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017YFC1310202
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Lingzhi; Traditional Chinese Medicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-start Group (Experimental): Receiving Lingzhi (Ganoderma in capsule form) 0.8g twice daily for 72 weeks
  Interventions: Drug: Ganoderma
- Delayed-start Group (Placebo Comparator): Receiving placebo for 24 weeks followed by Lingzhi (Ganoderma in capsule form) 0.8g twice daily for 48 weeks
  Interventions: Drug: Ganoderma; Drug: Placebos

INTERVENTIONS:
Drug: Ganoderma — 0.8g twice daily
  Other Names: Lingzhi
Drug: Placebos — 0.8g twice daily
  Arms: Delayed-start Group

SUMMARY:
Lingzhi(Ganoderma) is widely used in traditional Chinese medicine. Previous studies indicated that Lingzhi was safe, well tolorated, and improved symptoms as an add-on therapy to levodopa in early Parkinson's disease(PD) patients. Here the investigators design a multicenter, randomized, double-blind, placebo-controlled, delayed-start trial to evaluate the effects of Lingzhi on modifying disease progression in untreated PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the criteria for "Probable Parkinson's disease" according to 2015 MDS Clinical Diagnostic Criteria for Parkinson's Disease
* Aged 30-80 years
* Hoehn-Yahr Stage≤2
* UPDRS Part III subscores ranging from 10 to 30 points
* Disease duration of 5 years or less
* Untreated with antiparkinsonian drugs for at least two weeks preceding the trial
* Willing to sign the written informed consent

Exclusion Criteria:

* Atypical or secondary parkinsonism
* With psychiatric symptoms or a history of psychiatric diseases
* With cognitive impairment(MMSE score<24)
* Major liver or kidney dysfunction
* Participating in other clinical trials within 3 months preceding the current trial

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in UPDRS Part III subscores | 72 weeks
  Compare changes in UPDRS part III scores from baseline to week 72 between early-start group and delayed-start group
Changes in Schwab-England scores | 72 weeks
  Compare changes in Schwab-England scores from baseline to week 72 between early-start group and delayed-start group
Ratios of subjects in need of additional antiparkinsonian drugs | 72 weeks
  Compare ratios of subjects in need of additional antiparkinsonian drugs during the 72 week period between early-start group and delayed-start group

SECONDARY OUTCOMES:
Changes in ADAS-COG scores | 72 weeks
  Compare changes in ADAS-COG scores from baseline to week 72 between early-start group and delayed-start group

CONTACTS AND LOCATIONS:
Overall Officials: Erhe Xu, M.D., Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China